CLINICAL TRIAL: NCT05007483
Title: Efficacy of Diet on Quality of Life in Multiple Sclerosis
Acronym: EDQ
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Terry L. Wahls (Other)
Responsible Party: Sponsor-Investigator, Terry L. Wahls, Principle Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 202104639
Record Dates: First submitted 2021-08-09; First posted 2021-08-16 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: dietary; nutrition; fatigue; quality of life
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Fatigue | interventions — Eicosapentaenoic Acid; Docosahexaenoic Acids; Phosphatidylcholines; Diet, Ketogenic; Nutrition Policy

STUDY DESIGN:
Intervention Model Description: Randomized controlled study design
Who Masked: Investigator, Outcomes Assessor
Masking Description: Assessors and principle investigator masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Modified paleolithic elimination diet). (Experimental): Modified paleolithic elimination diet.
  Interventions: Dietary Supplement: BodyBio Balance Oil; Dietary Supplement: Kirunal Fish Oil; Dietary Supplement: BodyBio PC; Behavioral: Modified Paleolithic Elimination diet
- Group 2 (TROO) (Experimental): Time Restricted Olive Oil Based (TROO) Ketogenic Diet
  Interventions: Dietary Supplement: BodyBio Balance Oil; Dietary Supplement: Kirunal Fish Oil; Dietary Supplement: BodyBio PC; Behavioral: Time Restricted Olive Oil Based (TROO) Ketogenic Diet
- Group 3 Control (Active Comparator): Usual diet with Dietary Guidelines for Americans Diet information
  Interventions: Behavioral: Usual diet with Dietary Guidelines for Americans Diet information

INTERVENTIONS:
Dietary Supplement: BodyBio Balance Oil — nutraceutical supplement
  Other Names: 1400 mg linoleic acid/350 mg linolenic acid
  Arms: Group 1 (Modified paleolithic elimination diet).; Group 2 (TROO)
Dietary Supplement: Kirunal Fish Oil — nutraceutical supplement
  Other Names: 315 mg eicosapentanoic acid/ 105 mg docosahexaenoic acid
  Arms: Group 1 (Modified paleolithic elimination diet).; Group 2 (TROO)
Dietary Supplement: BodyBio PC — nutraceutical supplement
  Other Names: 1300 mg phosphatidylcholine
  Arms: Group 1 (Modified paleolithic elimination diet).; Group 2 (TROO)
Behavioral: Modified Paleolithic Elimination diet — 1. Complete elimination of all gluten-, dairy-, and egg-containing foods.
  2. Increase fruit and vegetable intake to 6-9 servings/day comprising of 2-3 servings each of the following categories: intensely colored, sulfur-rich, and leafy greens.
  3. Consume 6-12 ounces/day protein including organ meats and fatty fish.
  4. Consume fermented foods daily.
  5. Consume daily servings of algae, seaweed, and nutritional yeast.
  Arms: Group 1 (Modified paleolithic elimination diet).
Behavioral: Time Restricted Olive Oil Based (TROO) Ketogenic Diet — 1. Restriction of dietary carbohydrates to < 50 grams/day.
  2. Use olive oil (cold-pressed extra virgin preferred) to increase fat intake to >160 grams/day.
  3. Consume <100 grams/day protein.
  4. Limit dairy to 2 servings/day of whole fat options (completely exclude reduced fat dairy).
  5. Consume at least 3 servings/day non-starchy vegetables.
  Arms: Group 2 (TROO)
Behavioral: Usual diet with Dietary Guidelines for Americans Diet information — 1. Limit sodium to < 2,300 mg/day.
  2. Limit added sugar and saturated fat intake to <10% of kcal/day, respectively.
  3. Consume 5 servings of fruits and vegetables per day.
  4. Consume 6-9 ounce equivalents/day of grains, making at least half whole grain options.
  5. Consume 3 servings of reduced fat dairy per day.
  6. Consume 6 ounces/day protein foods.
  Arms: Group 3 Control

SUMMARY:
The overarching goal of this project is to critically evaluate the efficacy of incorporating dietary guidance within multiple sclerosis (MS) care for improving long-term quality of life (QoL) compared to usual care. The primary objective of this study is to evaluate the effect of two dietary interventions (time restricted olive oil based (TROO) ketogenic and modified Paleolithic elimination) on MS QoL compared to usual care control (Dietary Guidelines for America), and the secondary objectives and the long-term effects on, motor function, low-contrast vision sensitivity, fatigue, mood, and disease activity assessed by brain imaging.

DETAILED DESCRIPTION:
In the United States, MS affects nearly 1 million people with a 2.8:1 female to male ratio and the highest incidence rates among whites and African Americans. The economic cost of managing MS is substantial. In the U.S., the total medical costs for patients with MS increased from $116 million in 2002 to $198 million in 2013. MS is a chronic, neuroinflammatory, and neurodegenerative disease-causing symptoms of pain, fatigue, and changes in vision, cognition, and movement that greatly reduce quality of life (QoL) and the ability to maintain employment.

The overarching goal of this project is to critically evaluate the efficacy of incorporating dietary guidance within multiple sclerosis (MS) care for improving long-term quality of life (QoL) compared to usual care. The primary objective of this study is to evaluate the effect of two dietary interventions (time restricted olive oil based (TROO) ketogenic and modified Paleolithic elimination) on MS QoL compared to usual care control (Dietary Guidelines for America), and the secondary objectives and the long-term effects on, motor function, low-contrast vision sensitivity, fatigue, mood, and disease activity assessed by brain imaging.

The proposed study will consist of study participants attending 3 in-person site visits, months 0, 3, and 24, and online surveys every 3 months (months 0-24).

This study will use a randomized single-blind controlled design to test the short-term (6 months) and long-term (an additional 18 months) impact of the intervention diets on symptoms of MS including QoL and related outcomes stated above. We will use a fourteen-day run-in period to identify participants who are most likely to be successful in completing study procedures; this process has been effective in our previous studies. Participants who successfully complete all baseline self-reported outcomes and follow all study procedures during the seven-day run-in period will be scheduled for an on-site baseline visit for randomization to one of three diets (time restricted olive oil based (TROO) ketogenic and modified Paleolithic elimination and Dietary Guidelines for America).

On-site study visits will include blood draws, motor, cognitive, vision function assessments, and MRI. Motor assessments will include a 6-minute walk test, 25-foot walk test, 9-hole pegboard to test hand function, symbol digit exercise to test thinking functions, and critical flicker fusion test, ocular coherence tomography and low contrast vision sensitivity to test vision. The study participant will be escorted to the MRI unit to complete a non-contrast MRI of the brain. At the baseline visit, participants will be randomized. Participants assigned to the intervention diets will be given intervention specific educational materials including shopping lists, example menus and recipes, and the study supplements. Study participants randomized to the dietary guidelines for Americans diet will receive emails and/or text messages (approximately 3-6 weeks) to receive resources with websites for the Dietary Guidelines of America, and recent multiple sclerosis-related research that does not involve diet.

Study team will provide fish oil, essential fatty acids, and phosphatidylcholine to the two intervention groups only. The participant will be scheduled for a Zoom video conference meeting with the assigned registered dietitian to review the assigned study diet.

In addition, subjects will collect saliva specimens for microbiome analysis at each of the 3 site study visits (months 0, 3 and 24).

Dietary History Questionnaire III will be completed at months 0, 3, 12 and 24 and will be used to assess adherence to the assigned dietary pattern.

The online questionnaires sent to participants every 3 months will also be used to track supplement intake, medication use, and details about health & life events, MS symptoms, fatigue, quality of life, doctor's appointment, and side effects they may be experiencing.

ELIGIBILITY:
Eligibility for the run-in phase of the study:

Participants will be eligible to enroll in the fourteen-day run-in phase of the study if they meet the following inclusion and exclusion criteria:

INCLUSION CRITERIA:

* A definitive diagnosis of RRMS based on the 2017 revised McDonald Criteria.
* The ability to prepare, or availability of someone to prepare, home-cooked meals.
* Must own a computer, smartphone, or tablet device that has internet access to complete online surveys and capable of running study related applications.
* Must be willing to follow study procedures outlined and explained to them.
* Be between the ages of 18 to 70 at the time of consent.
* Must be able to walk 25 feet without support.
* Willingness to be randomized and follow any of the study diets.
* Must consent to sharing the clinical notes from their primary care and neurology providers during the study period.

EXCLUSION CRITERIA:

* Moderate or severe mental impairment.
* Use of insulin, Coumadin, weight loss medications such as orlistat that causes fat malabsorption.
* Worsening of symptoms resulting in the initiation or change of treatment including steroids (solumedrol, prednisone, etc.) or disease-modifying medications in 4 weeks prior to consent.
* Treatment for cancer by radiation or chemotherapy in 12 months prior to consent, other than skin cancer.
* Diagnosis of clinically significant heart disease, liver disease, kidney disease, or history of oxalate kidney stones.
* Diagnosis of type II diabetes that does not have approval from treating physicians to adopt any of the 3 study diets.
* Clinical diagnosis of moderate to severe psychiatric disease that makes study adherence more difficult (e.g., schizophrenia, bi-polar disease, severe depression and/or anxiety).
* An active eating disorder such as anorexia, bulimia, binge eating, or orthorexia.
* Measurement of BMI <20.
* Confirmation of pregnancy or planning to become pregnant in the next 2 years.
* History of diagnosed fat intolerance/malabsorption such as cholecystectomy or uncontrolled exocrine pancreatic insufficiency.
* Participation in another research study investigating MS treatments, diet, or exercise.
* Presence of a contraindication to completing a brain MRI or having claustrophobia which interferes with completion of MRI studies without the use of sedation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Multiple Sclerosis 54 Quality of Life Mental Health (MS 54 QoL MH) | baseline to 3 Months
  Change in (MS 54 QoL MH) survey questions mean scores, range 0-100, higher number is better.
Multiple Sclerosis 54 Quality of Life Mental Health (MS 54 QoL MH) | baseline to 6 Months
  Change in (MS 54 QoL MH) survey questions mean scores, range 0-100, higher number is better.
Multiple Sclerosis 54 Quality of Life Mental Health (MS 54 QoL MH) | baseline to 12 Months
  Change in (MS 54 QoL MH) survey questions mean scores, range 0-100, higher number is better.
Multiple Sclerosis 54 Quality of Life Mental Health (MS 54 QoL MH) | baseline to 18 Months
  Change in (MS 54 QoL MH) survey questions mean scores, range 0-100, higher number is better.
Multiple Sclerosis 54 Quality of Life Mental Health (MS 54 QoL MH) | baseline to 24 Months
  Change in (MS 54 QoL MH) survey questions mean scores, range 0-100, higher number is better.
Multiple Sclerosis 54 Quality of Life Physical Health (MS 54 QoL PH) | baseline to 3 Months
  Change in (MS 54 QoL PH) survey questions mean scores, range 0-100, higher number is better.
Multiple Sclerosis 54 Quality of Life Physical Health (MS 54 QoL PH) | baseline to 6 Months
  Change in (MS 54 QoL PH) survey questions mean scores, range 0-100, higher number is better.

SECONDARY OUTCOMES:
Modified Fatigue Impact Scale (MFIS) | baseline to 3 months
  Change in MFIS survey questions, scores range from 0-84, lower score is better.
Modified Fatigue Impact Scale (MFIS) | baseline to 6 months
  Change in MFIS survey questions, scores range from 0-84, lower score is better.
Modified Fatigue Impact Scale (MFIS) | baseline to 12 months
  Change in MFIS survey questions, scores range from 0-84, lower score is better.
Modified Fatigue Impact Scale (MFIS) | baseline to 18 months
  Change in MFIS survey questions, scores range from 0-84, lower score is better.
Modified Fatigue Impact Scale (MFIS) | baseline to 24 months
  Change in MFIS survey questions, scores range from 0-84, lower score is better.
Hospital Anxiety Depression Scale (HADS) | baseline to 3 months
  Change in HADS survey question score, a 14 question scale ranging from 0-3 with zero being being low or no occurrence and 3 being high occurrence
Hospital Anxiety Depression Scale (HADS) | baseline to 6 months
  Change in HADS survey question score, a 14 question scale ranging from 0-3 with zero being being low or no occurrence and 3 being high occurrence
Hospital Anxiety Depression Scale (HADS) | baseline to 12 months
  Change in HADS survey question score, a 14 question scale ranging from 0-3 with zero being being low or no occurrence and 3 being high occurrence
Hospital Anxiety Depression Scale (HADS) | baseline to 18 months
  Change in HADS survey question score, a 14 question scale ranging from 0-3 with zero being being low or no occurrence and 3 being high occurrence
Hospital Anxiety Depression Scale (HADS) | baseline to 24 months
  Change in HADS survey question score, a 14 question scale ranging from 0-3 with zero being being low or no occurrence and 3 being high occurrence
Fatigue Severity Scale score (FSS) | Baseline to 3 months
  Change in FSS survey question mean scores, scores range from 1-7, lower is better.
Fatigue Severity Scale score (FSS) | Baseline to 6 months
  Change in FSS survey question mean scores, scores range from 1-7, lower is better.
Fatigue Severity Scale score (FSS) | Baseline to 12 months
  Change in FSS survey question mean scores, scores range from 1-7, lower is better.
Fatigue Severity Scale score (FSS) | Baseline to 18 months
  Change in FSS survey question mean scores, scores range from 1-7, lower is better.
Fatigue Severity Scale score (FSS) | Baseline to 24 months
  Change in FSS survey question mean scores, scores range from 1-7, lower is better.
Brain volume as measured by non contrast magnetic resonance imaging (MRI) | baseline to 24 months
  Change in MRI grey matter brain volume, more is better
Brain lesions as measured by non contrast magnetic resonance imaging (MRI) | baseline to 24 months
  Change in inflammatory lesions numbers as measured by non contrast brain MRI, fewer is better
Timed 25 foot walk test | baseline to 3 months
  seconds required to walk 25 feet, lower is better
Timed 25 foot walk test | baseline to 24 months
  seconds required to walk 25 feet, lower is better
9 Hole peg board test | baseline to 3 months
  seconds require to move 9 pegs to various locations on a peg board, fewer seconds is better
9 Hole peg board test | baseline to 24 months
  seconds require to move 9 pegs to various locations on a peg board, fewer seconds is better
Low contrast visual acuity | baseline to 3 months
  A measure of best corrected vision, measure is log minimal angle of resolution at 2.5% contrast. Lower number is better.
Low contrast visual acuity | baseline to 24 months
  A measure of best corrected vision, measure is log minimal angle of resolution at 2.5% contrast. Lower number is better.
Dietary History Questionnaire IIi | baseline to 12 months
  Change in dietary intake measured by survey questions
Dietary History Questionnaire IIi | baseline to 3 months
  Change in dietary intake measured by survey questions
Critical flicker fusion | baseline to 3 months
  change in The herz at which a flickering light is seen as non-flickering as measured by herz
Critical flicker fusion | baseline to 24 months
  change in The herz at which a flickering light is seen as non-flickering as measured by herz
Ocular Coherence tomography | baseline
  Measure of optic nerve and retina depths using infrared light technology
Ocular Coherence tomography | baseline to 3 months
  change in the Measure of optic nerve and retina depths using infrared light technology
Ocular Coherence tomography | baseline to 24 months
  change in the Measure of optic nerve and retina depths using infrared light technology
Neurofilament light chain | baseline to 3 months
  blood biomarker of neuroaxonal (brain) damage
Neurofilament light chain | baseline to 24 months
  blood biomarker of neuroaxonal (brain) damage
Multiple Sclerosis 54 Quality of Life Physical Health (MS 54 QoL PH) | baseline to 12 Months
  Change in (MS 54 QoL PH) survey questions mean scores, range 0-100, higher number is better.
Multiple Sclerosis 54 Quality of Life Physical Health (MS 54 QoL PH) | baseline to 18 Months
  Change in (MS 54 QoL PH) survey questions mean scores, range 0-100, higher number is better.
Multiple Sclerosis 54 Quality of Life Physical Health (MS 54 QoL PH) | baseline to 24 Months
  Change in (MS 54 QoL PH) survey questions mean scores, range 0-100, higher number is better.

CONTACTS AND LOCATIONS:
Overall Officials: Terry L Wahls, MD, Principal Investigator — University of Iowa
Locations (1):
- Univeristy of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wahls TL, Chenard CA, Snetselaar LG. Review of Two Popular Eating Plans within the Multiple Sclerosis Community: Low Saturated Fat and Modified Paleolithic. Nutrients. 2019 Feb 7;11(2):352. doi: 10.3390/nu11020352. PMID 30736445
- [Result] Wahls T, Scott MO, Alshare Z, Rubenstein L, Darling W, Carr L, Smith K, Chenard CA, LaRocca N, Snetselaar L. Dietary approaches to treat MS-related fatigue: comparing the modified Paleolithic (Wahls Elimination) and low saturated fat (Swank) diets on perceived fatigue in persons with relapsing-remitting multiple sclerosis: study protocol for a randomized controlled trial. Trials. 2018 Jun 4;19(1):309. doi: 10.1186/s13063-018-2680-x. PMID 29866196
- [Result] Chenard CA, Rubenstein LM, Snetselaar LG, Wahls TL. Nutrient Composition Comparison between a Modified Paleolithic Diet for Multiple Sclerosis and the Recommended Healthy U.S.-Style Eating Pattern. Nutrients. 2019 Mar 1;11(3):537. doi: 10.3390/nu11030537. PMID 30832289
- [Result] Titcomb TJ, Bisht B, Moore DD 3rd, Chhonker YS, Murry DJ, Snetselaar LG, Wahls TL. Eating Pattern and Nutritional Risks among People with Multiple Sclerosis Following a Modified Paleolithic Diet. Nutrients. 2020 Jun 20;12(6):1844. doi: 10.3390/nu12061844. PMID 32575774
- [Result] Lee JE, Bisht B, Hall MJ, Rubenstein LM, Louison R, Klein DT, Wahls TL. A Multimodal, Nonpharmacologic Intervention Improves Mood and Cognitive Function in People with Multiple Sclerosis. J Am Coll Nutr. 2017 Mar-Apr;36(3):150-168. doi: 10.1080/07315724.2016.1255160. Epub 2017 Apr 10. PMID 28394724
- [Result] Lee JE, Titcomb TJ, Bisht B, Rubenstein LM, Louison R, Wahls TL. A Modified MCT-Based Ketogenic Diet Increases Plasma beta-Hydroxybutyrate but Has Less Effect on Fatigue and Quality of Life in People with Multiple Sclerosis Compared to a Modified Paleolithic Diet: A Waitlist-Controlled, Randomized Pilot Study. J Am Coll Nutr. 2021 Jan;40(1):13-25. doi: 10.1080/07315724.2020.1734988. Epub 2020 Mar 26. PMID 32213121
- [Result] Chenard CA, Rubenstein LM, Snetselaar LG, Wahls TL. Nutrient Composition Comparison between the Low Saturated Fat Swank Diet for Multiple Sclerosis and Healthy U.S.-Style Eating Pattern. Nutrients. 2019 Mar 13;11(3):616. doi: 10.3390/nu11030616. PMID 30871265
- [Result] Irish AK, Erickson CM, Wahls TL, Snetselaar LG, Darling WG. Randomized control trial evaluation of a modified Paleolithic dietary intervention in the treatment of relapsing-remitting multiple sclerosis: a pilot study. Degener Neurol Neuromuscul Dis. 2017 Jan 4;7:1-18. doi: 10.2147/DNND.S116949. eCollection 2017. PMID 30050374
- [Result] Bisht B, Darling WG, Grossmann RE, Shivapour ET, Lutgendorf SK, Snetselaar LG, Hall MJ, Zimmerman MB, Wahls TL. A multimodal intervention for patients with secondary progressive multiple sclerosis: feasibility and effect on fatigue. J Altern Complement Med. 2014 May;20(5):347-55. doi: 10.1089/acm.2013.0188. Epub 2014 Jan 29. PMID 24476345
- [Derived] Shemirani F, Klein AM, Groux AR, Kilpatrick R, Brooks L, Ehlinger MA, Darling WG, Magnotta VA, Gill CM, Hoth KF, Mangalam A, Eyck PT, Martinez AS, Hook J, Titcomb TJ, Snetselaar LG, Wahls TL. Efficacy of Diet on Quality of life in Multiple Sclerosis (EDQ-MS): a study protocol for a randomized controlled clinical trial. Trials. 2025 Oct 27;26(1):437. doi: 10.1186/s13063-025-09157-2. PMID 41146285